CLINICAL TRIAL: NCT02818374
Title: Evaluation of the Efficacy and Safety of Use of an Innovative Medical Device for Improving Oral Accessibility in People With Disabilities, Presenting Behavioral Disorders: The Oral Accessibility Spatula (Spatule SAB)
Brief Title: The Oral Accessibility Spatula (Spatule SAB)
Acronym: SAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-02-CHRMT
Record Dates: First submitted 2016-03-30; First posted 2016-06-29 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-02

CONDITIONS: Mental Handicap
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disabled People with behavioral trouble (Experimental)
  Interventions: Device: oral accessibility spatula (SAB)

INTERVENTIONS:
Device: oral accessibility spatula (SAB)

SUMMARY:
The purpose of this study is to evaluate the efficiency and the safe use of a new medical device to improve the oral accessibility of disabled people during the oral-dental examination.

DETAILED DESCRIPTION:
The oral examination of people with behavioural handicap seems to be difficult. Those patients react with defensive reflexes which limit spontaneously the amplitude of their oral cavity or prevent them to keep open their mouth for a sufficient time to process the examination. This difficulty can be caused by various reasons: cerebral motor disability, behavioral troubles or mental disability, and it affects people of all ages.

The current methods keeping open the mouth like wedges are often unsuitable for those patients. Moreover, no other device exists or is described even in literature. An innovative medical device has to be developed, in order to offer to disabled patients and the users or dentists a comfort during the oral-dental examination.

The oral accessibility spatula, made out polypropylene plastic, is designed into two parts :

* a handle to hold the spatula by the user
* a thin plastic surface introduced into the mouth, which is dull with a round edge and has holes on the sides to lock the spatula between the upper and lower teeth.

Primary objective :

To evaluate the buccal access during a first oral-dental examination without and then with the oral accessibility spatula (SAB).

Secondary objective :

To evaluate the safe use of the SAB To evaluate the tolerance of the exam without, and then with the SAB

Primary endpoint :

Visibility and dental examination of incisor-canine sectors, premolars and molars using a probe, assessed by an oral accessibility score determined based on intra oral accessible areas with and without oral accessibility Spatula device

Secondary endpoints :

The safety of the spatula will be assessed by analyzing the reported adverse effects and their relative frequency The dental exam tolerance evaluation; with and without Oral Accessibility .Spatula

Methodology :

Multi-center interventional prospective study, open-label Only one medical check per patient

Procedures :

Any patient with a behavioral handicap, and who consults with dentist for a preventive check-up or a oral-dental curative act, is examined by an inclusion operator who checks the inclusion or non-inclusion criteria, and especially the behavior with Venham Scale (only patients with a score of 2 and higher, meaning opposing, after an approach toward the oral cavity are included).

The oral accessibility score of each eligible patient is performed twice, without the SAB first, and then with the SAB.

The incidents and/or potential injuries are reported from a standardized grid. Venham scale score is measured a second time during the oral-dental examination without or with the spatula.

Patients number :

Without the SAB, the rate of patients with an oral accessibility score of at least level 8 is 20%.

The protocol forecasts hypothetically a 20% highering of this rate after the use of SAB (so 40% of patients with a score of 8 and higher). With a total staff of 140 patients, this hypothesis is validated with an α risk set at 5% and a statistical power at 90%. 200 patients are expected in order to take into account a potential center effect and a potential investigator effect, and a study output rate of 10%.

Trial Time :

Only one medical check per patient, so the total duration goes with the inclusion period of 18 months.

Expected study start : first semester of 2016 End of inclusion : second semester of 2017 End of study : second semester of 2017

Statistical Analysis :

The major analysis will be the comparison of the oral accessibility scores during the examination with or without the SAB. Each patient will be his own control, and the examinations always will be performed without the SAB in first, and secondly with the SAB, by the same dental surgeon.

Expected Benefits :

The expected result is the proof of a best examination quality with no risk for the patient. The major prospect is the availability of the SAB to dental surgeons to improve the therapeutic indications and the quality of examinations, then to parents, carers and caregivers, in order to make possible and easier the application of a oral-dental health suitable for handicapped or disabled people.

So, the expected benefits are :

* early diagnostic of the oral-dental diseases
* improved efficiency of the tooth care
* reduction of the use of general anesthesia for oral examinations
* help for tooth washing in order to improve significantly the oral-dental healthy level
* improved prevention by the availability of the spatula to parents, carers and physicians.

Quality Assurance Plan :

Data will be recorded in a Paper Case Report from medical records. The patients will undergo only one medical examination for the study. No follow-up is expected.

ELIGIBILITY:
Inclusion Criteria:

* Mental disability patient with behavioural troubles known or noticed during the approach of hand for dental examination
* Venham Scale score of 2 and higher, meaning opposing, after an approach toward the oral cavity
* Information of the responsible person for the patient, if necessary, and followed by the dated signed informed consent

Exclusion Criteria:

* pregnant or nursing woman
* lack of social security
* people under guardianship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Visibility and dental examination of incisor-canine sectors, premolars and molars using a probe, assessed by an oral accessibility score determined based on intra oral accessible areas with and without oral accessibility Spatula device | 1 day
  score of 0 = no access to 12 = total accessibility

SECONDARY OUTCOMES:
The safety of the spatula will be assessed by analyzing the reported adverse effects and their relative frequency | 1 day
The dental exam tolerance evaluation with and without Oral Accessibility Spatula | 1 day
  using Venham behaviour scale

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Dijon, Dijon
  - Centre Hospitalier Emile Durkheim, Épinal
  - Clinique Saint Francois, Haguenau
  - CHR Metz-Thionville- Mercy Hospital, Metz
  - CHRU Nancy, Nancy
  - CHRU Strasbourg, Strasbourg
  - CHR METZ THIONVILLE- Bel-Air Hospital, Thionville

IPD SHARING:
Plan to Share IPD: No